CLINICAL TRIAL: NCT00432653
Title: Open Label Clinical Trial With Rituximab (MabThera ®) in Ankylosing Spondylitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ritux-AS-01
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2007-02-08 (Estimated); Status verified 2007-02

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; rituximab; therapy; magnetic resonance imaging
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
To evaluate the efficacy and safety of rituximab when added to NSAIDs and/ or methotrexate both for TNFalpha inhibitor naïve or TNFalpha inhibitor failure patients with moderate to severe ankylosing spondylitis

DETAILED DESCRIPTION:
Indication: Moderate to severe ankylosing spondylitis who have had an inadequate response to or do not tolerate conventional therapy including NSAIDs, DMARDs and TNF alpha inhibitors.

Rationale: We have argued already 10 years ago that autoimmunity plays an important role in the pathogenesis of ankylosing spondylitis (AS). Although there is no direct evidence, as in nearly all 'suspected' autoimmune diseases, of an autoimmune response in AS it has been proposed repeatedly over the last years that the cartilage is the most likely target of an autoimmune response in AS. Histological studies 4,5 and magnet resonance imaging investigations suggest that the primary site of inflammation is the cartilage/bone interphase. Mononuclear cell infiltrates are mainly found in cartilage and the subchondral bone. In early and active sacroiliitis, T cells and macrophages are dominant in these infiltrates underlining the relevance of a specific cellular immune response 5.Furthermore, T cell responses have been demonstrated against proteoglycan (an important cartilage protein) in human arthritides including ankylosing spondylitis. We could also recently demonstrate both a CD4+ and a CD8+ T cell response to proteogkycan (aggrecan) derived peptides in the peripheral blood and a CD8+ T cell response against a collagen VI derived peptide in the synovial fluid from AS patients. Thus, all these findings suggest that a chronic, probably T cell mediated, immune response against cartilage is relevant in the pathogenesis of AS.This was further backed by recent studies from our group demonstrating mononuclear infiltrates of cartilage by investigating femoral heads and facette joints (small joints of the spine) obtained by surgery from a number of AS patients). The presence of mononuclear cell infiltrates was strongly dependent on the presence of cartilage on the surface of the femoral heads, suggesting that cartilage could be indeed the stimulus and target of a cellular immune response. However, rather surprisingly there were also dense infiltrations of B cells in the subchondral bone marrow in these patients. In comparison to immunohistological stainings from controls without spinal disease, the number of B cells in AS was even higher than the T cells. At the moment it is not clear whether this indicates that autoantibodies do play a role in the pathogenesis or whether these B cells might rather act as important local antigen presenting cells. In any case, given the assumed autoimmune pathogenesis in AS and the presence of B cells aggregates in inflammatory cellular infiltrates the study of potential effects of an immunotherapy which targets B cells in AS is justified and needed.

Objectives: To evaluate the efficacy and safety of rituximab when added to NSAIDs and/ or methotrexate both for TNFalpha inhibitor naïve or TNFalpha inhibitor failure patients with moderate to severe ankylosing spondylitis.

Study design: Open label clinical trial with a study duration of 48 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 65 years of age who have moderate to severe ankylosing spondylitis.
* Active disease is defined as a BASDAI score of ³ 4 plus a
* back pain score (BASDAI question 2) of ³ 4 despite concurrent NSAID therapy, or intolerance to NSAIDs
* If on prednisone, £10 mg per day must be stable for 4 weeks prior to baseline.
* If on methotrexate, £ 25 mg per week must be stable for 4 weeks prior to baseline
* If on sulfasalazine, must be stable 4 weeks prior to basline
* Women of child bearing potential must have a negative pregnancy urine test at study baseline and use an adequate, effective method of contraception (such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence, vasectomised partner) for a duration of 12 months after stop of rituximab therapy.
* Sexual active men must use an accepted method of contraception for a duration of 12 months after first administration of rituximab.
* Willingness and capability to give written informed consent, written consent for data protection (legal requirement in Germany: datenschutzrechtliche Einwilligung) and willingness to participate and to comply with the study

Exclusion Criteria:

Exclusion criteria related to general health conditions

* Patients with other chronic inflammatory articular disease or systemic autoimmune disease, e.g. Systemic lupus erythematosus,Sjögren's syndrome, active rheumatoid vasculitis, a history of systemic diseases associated with arthritis, chronic fatigue syndrome
* Any active infection, a history of recurrent clinically significant infection, a history of recurrent bacterial infections with encapsulated organisms
* Primary or secondary immunodeficiency
* History of cancer with curative treatment not longer than 5 years ago except basal-cell carcinoma of the skin that had been excised
* A history of pulmonary or cardiac insufficiency, or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease ( e.g. heart failure class III/IV NYHA, cardiac infarct within last 6 month), nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders.
* Neuropathy that can interfere with quality of life and/or pain assessment.
* Patients with a history of a severe psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
* History of current evidence of abuse of "hard" drugs (e.g. cocaine/ heroine) or alcoholism
* Known hypersensitivity to any component of the product or to murine proteins (sodium citrate, polysorbate 80, sodium chloride, sodium hydroxide, HCl).
* Women lactating, pregnant, nursing or of childbearing potential with a positive pregnancy test (urine test)
* Males or females of reproductive potential not willing to use effective contraception (e.g. contraceptive pill, IUD, physical barrier) for up to 12.5 months after first infusion of rituximab
* History of alcohol, drug or chemical abuse within 6 month prior to screening
* Lack of peripheral venous access

Exclusion criteria related to medications

* Obligatory indication for initiation of established therapy, e.g. with TNFalpha-inhibitors
* If on leflunomide, leflunomide must have been terminated at least 8 weeks prior to the first rituximab infusion (or ≥ 28 days after 11 days of standard cholestyramine or activated charcoal washout).
* If on TNFalpha blocking agent (infliximab, etancercept, adalimumab), the TNFa therapy must have been terminated at least 4 weeks prior to the first rituximab infusion if etanercept was used and at least 8 weeks if infliximab or adalimumab were used
* Previous treatment with rituximab or intolerance to rituximab
* Corticosteroids at doses exceeding 10 mg per day of prednisolone or the equivalent within the last 4 weeks prior to the first rituximab infusion
* Intolerance or contraindication to drugs required for the treatment of the side effects of rituximab (e.g. paracetamol, acetaminophen, diphenhydramine, p.o. and i.v. corticosteroids, anti-emetics or H1 blockers
* Previous treatment with any investigational agent
* Previous treatment with i.v. immunoglobulins
* Receipt of a live vaccine within 4 weeks prior to treatment
* Intra-articular or parenteral corticosteroids within 4 weeks prior to screening visit

Exclusion criteria related to lab findings

* Haemoglobin < 8.5 g/dl
* Neutrophil counts < 2.000 / µl
* Platelet count < 125.000 / µl
* Lower than 1 x 1000/µl lymphopenia for more than three months prior to inclusion.
* Serum creatinine > 1.4 mg/dl for women or 1.6 mg/dl for men.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times upper limit of normal
* Positive HIV, hepatitis B or C serology

Exclusion criteria related to formal aspects

* Patients who participate currently in another clinical trial or patients who participated in another clinical trial during the last 30 days.
* Patients who are underage or patients who are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to § 40 Abs. 4 and § 41 Abs. 2 und Abs. 3 AMG).
* Patients who are institutionalised due to regulatory or juridical order (according to AMG § 40 (1) Abs. 4)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2007-03; Study Completion 2009-11

PRIMARY OUTCOMES:
Evaluation in week 24 and until study end: ASAS 20 in AS patients naïve to TNFalpha inhibitors as well as in AS patients with previous therapy with TNFalpha inhibitors.

SECONDARY OUTCOMES:
Safety Evaluations (Adverse events, vital signs, physical examination results, and clinical laboratory values until week 48)
Efficacy Evaluations:
ASAS 40 response
ASAS criteria for partial remission
Duration of response
BASDAI 20%, 50%, 70% improvement
BASFI
Mobility examinations
BASMI
Chest Wall Expansion
disease controlling antirheumatic therapy criteria (DC-ART20) (5 out of 6)
CRP, ESR
Quality of Life
SF-36Numeric Rating Scale (NRS)
physicians global
patients global
general pain
nocturnal pain Enthesitis index (Maastricht scale
swollen joint countEQ-5D
Socio-economic questionnairecourse of change of active and chronic inflammatory lesions in MRI after 24 weeks and after 48 weeksB cell analysis and T cell analysis

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, MD, Prof., Principal Investigator — Charite, Campus Benjamin-Franklin, Med. Clinic I, Rheumatology, Hindenburgdamm 30, 12200 Berlin, Germany
Locations (2):
- Germany (2):
  - Charite, Campus Benjamin-Franklin, Med. Clinic I, Rheumatology, Berlin
  - Rheumazentrum Ruhrgebiet, St. Josefs Krankenhaus, Herne

REFERENCES:
- [Background] Sieper J, Braun J. Pathogenesis of spondylarthropathies. Persistent bacterial antigen, autoimmunity, or both? Arthritis Rheum. 1995 Nov;38(11):1547-54. doi: 10.1002/art.1780381105. PMID 7488274
- [Background] Appel H, Loddenkemper C, Grozdanovic Z, Ebhardt H, Dreimann M, Hempfing A, Stein H, Metz-Stavenhagen P, Rudwaleit M, Sieper J. Correlation of histopathological findings and magnetic resonance imaging in the spine of patients with ankylosing spondylitis. Arthritis Res Ther. 2006;8(5):R143. doi: 10.1186/ar2035. PMID 16925803
- [Background] Appel H, Kuhne M, Spiekermann S, Ebhardt H, Grozdanovic Z, Kohler D, Dreimann M, Hempfing A, Rudwaleit M, Stein H, Metz-Stavenhagen P, Sieper J, Loddenkemper C. Immunohistologic analysis of zygapophyseal joints in patients with ankylosing spondylitis. Arthritis Rheum. 2006 Sep;54(9):2845-51. doi: 10.1002/art.22060. PMID 16947385
- [Background] Zochling J, van der Heijde D, Burgos-Vargas R, Collantes E, Davis JC Jr, Dijkmans B, Dougados M, Geher P, Inman RD, Khan MA, Kvien TK, Leirisalo-Repo M, Olivieri I, Pavelka K, Sieper J, Stucki G, Sturrock RD, van der Linden S, Wendling D, Bohm H, van Royen BJ, Braun J; 'ASsessment in AS' international working group; European League Against Rheumatism. ASAS/EULAR recommendations for the management of ankylosing spondylitis. Ann Rheum Dis. 2006 Apr;65(4):442-52. doi: 10.1136/ard.2005.041137. Epub 2005 Aug 26. PMID 16126791
- [Background] Edwards JC, Szczepanski L, Szechinski J, Filipowicz-Sosnowska A, Emery P, Close DR, Stevens RM, Shaw T. Efficacy of B-cell-targeted therapy with rituximab in patients with rheumatoid arthritis. N Engl J Med. 2004 Jun 17;350(25):2572-81. doi: 10.1056/NEJMoa032534. PMID 15201414
- [Background] Emery P, Fleischmann R, Filipowicz-Sosnowska A, Schechtman J, Szczepanski L, Kavanaugh A, Racewicz AJ, van Vollenhoven RF, Li NF, Agarwal S, Hessey EW, Shaw TM; DANCER Study Group. The efficacy and safety of rituximab in patients with active rheumatoid arthritis despite methotrexate treatment: results of a phase IIB randomized, double-blind, placebo-controlled, dose-ranging trial. Arthritis Rheum. 2006 May;54(5):1390-400. doi: 10.1002/art.21778. PMID 16649186
- [Background] Sieper J, Baraliakos X, Listing J, Brandt J, Haibel H, Rudwaleit M, Braun J. Persistent reduction of spinal inflammation as assessed by magnetic resonance imaging in patients with ankylosing spondylitis after 2 yrs of treatment with the anti-tumour necrosis factor agent infliximab. Rheumatology (Oxford). 2005 Dec;44(12):1525-30. doi: 10.1093/rheumatology/kei046. Epub 2005 Aug 9. PMID 16091396
- [Derived] Song IH, Heldmann F, Rudwaleit M, Listing J, Appel H, Braun J, Sieper J. Different response to rituximab in tumor necrosis factor blocker-naive patients with active ankylosing spondylitis and in patients in whom tumor necrosis factor blockers have failed: a twenty-four-week clinical trial. Arthritis Rheum. 2010 May;62(5):1290-7. doi: 10.1002/art.27383. PMID 20461780